CLINICAL TRIAL: NCT03783390
Title: Brain, Activity, Teens, and Exercise (BATE)
Brief Title: Brain, Appetite, Teens, and Exercise
Acronym: BATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Robin Shook, Research Faculty PhD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00000096
Record Dates: First submitted 2018-07-17; First posted 2018-12-21 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Energy Balance; Appetitive Behavior; Obesity
MeSH Terms: conditions — Appetitive Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: To assess the effectiveness of a physical activity intervention on eating behavior in adolescents; OW/OB inactive adolescents will be randomly assigned to a 3-month exercise intervention (Exercise +Newsletter), or a control condition (Newsletter).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Orientation (No Intervention): Informed consent, height, weight, and blood pressure measurement. A link to an online survey the participant and their parent can fill out at home about the participant's medical history will be given.
- Measurement session Pre/Post Intervention (No Intervention): Questionnaires completed, blood draws, and fixed and ad lib meals completed to measure appetite and hormones. DXA completed.
- Home Assessments Pre/Post intervention (No Intervention): 24-hour dietary recalls. Physical activity measured by monitors (Actigraph, ActivPAL).
- Physical Activity Session Pre/Post intervention (No Intervention): DXA, and Fitness testing to measure VO2submax and VO2max. Cognitive assessments will be administered.
- fMRI Session Pre/Post intervention (No Intervention): The participant will have an fMRI completed and answer questions related to 60 food and activity images while in and out of the fMRI machine.
- Exercise Intervention/Newsletter (Experimental): After completion of the initial fMRI session the participant will be randomly assigned to intervention for 3 months and then complete another round of assessments described as above (except for the orientation session).
  Interventions: Behavioral: Exercise Intervention; Behavioral: Newsletter

INTERVENTIONS:
Behavioral: Exercise Intervention — Youth randomized to the active condition will participate in an organized exercise program. During the exercise program, adolescents will participate in a supervised structured exercise (treadmill walking/cycling on stationary bike) on 3 days equivalent to approximately 180 min/week of moderate-intensity exercise. The rationale for this dose of structured exercise is based on national (ADA) and international physical activity recommendations for youth of 60 minutes/day.
  Arms: Exercise Intervention/Newsletter
Behavioral: Newsletter — Families will receive a monthly newsletter with "parenting tips, sample praise statements, and child-appropriate activities and recipes" identical to what has been used in the work of leaders in the field of pediatric obesity. Previous research suggests that newsletter/mail interventions are well received by participants and are frequently included in federally funded health intervention studies.
  Arms: Exercise Intervention/Newsletter

SUMMARY:
The long-term goal is to develop effective, evidence-based lifestyle interventions to prevent and treat childhood obesity and related co-morbidities. The short-term goal, and the purpose of this application, is to quantify appetite and neural mechanisms of food reward in overweight/obese (OW/OB) sedentary youth and to quantify changes following the implementation of a physical activity intervention. The central hypothesis is that appetite becomes dysregulated at low levels of physical activity via neural reward pathways, and appetite control will improve following a long-term exercise intervention. The investigators consider this project a pilot study designed to generate data to be used for future external funding opportunities, demonstrate collaboration between researchers, and test the feasibility of the protocols.

DETAILED DESCRIPTION:
Specific Aim 1: To identify associations between neural, psychological, and hormonal appetite control pathways using subjective and objective measures of appetite and neurocognitive assessments of reward pre-intervention.

Hypothesis 1: There will be significant cross-modulation of appetite across neural (brain activation), psychological (subjective hunger), and hormonal pathways (satiety biomarkers), though the temporal relationship between each in response to feeding is unknown.

Specific Aim 2: To assess the effectiveness of a physical activity intervention on eating behavior in adolescents; OW/OB inactive adolescents will be randomly assigned to a 3-month exercise intervention (Exercise +Newsletter), or a control condition (Newsletter).

Hypothesis 2a: Those exposed to the exercise intervention will have greater improvements (compared to control group) in appetite (subjective self-reported hunger and palatability responses, and, objectively, satiety and appetite hormones glucose, insulin, ghrelin, and leptin, and calories consumed during ad libitum meal).

Hypothesis 2B. Compared to pre-intervention, OB/OW youth in the exercise group will show decreased reward activation in regions of the brain when making decisions about appetizing foods compared to post-intervention when hungry and when fed. In self-control regions, compared to pre-intervention, the investigators will observe increased activity in both hungry and fed conditions.

At the end of the proposed study, it is the expectation that the investigators will have collected important preliminary data regarding how long-term structured exercise acts upon appetite and neural mechanisms related to food reward in adolescents. Findings are key not only to interventions targeting OW/OB youth, but also to public policy and health recommendations for the importance of physical activity in children.

ELIGIBILITY:
Inclusion Criteria

* Overweight/obese (BMI ≥85th to <99th percentile for age and sex)
* Weight stable
* Ages 14-17
* No meds that may alter metabolism
* Sedentary (<20 min/day exercise)
* At risk for T2D, according to American Diabetes Association (ADA) criteria:

  * family history of T2D in first- or second- degree relative
  * Race/ethnicity (Native American, African American, Latino, Asian American, Pacific Islander)
  * Signs of insulin resistance
  * Maternal history of diabetes for gestational diabetes during child's gestation
* Willing to participate in an exercise program
* Willing to provide permission/assent

Exclusion Criteria:

* BMI <85th percentile for age and sex
* Weight not stable
* Age <14 or >17
* On meds that may alter metabolism
* Active (>20 min/day exercise)
* Not at risk for T2D, according to American Diabetes Association (ADA) criteria (see above)
* Not willing to participate in an exercise program
* Not willing to provide permission/assent

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Assess the effectiveness of a physical activity intervention on eating behavior- subjective responses | 12 monthts
  To assess the effectiveness of a physical activity intervention on eating behavior in adolescents; OW/OB inactive adolescents will be randomly assigned to a 3-month exercise intervention (Exercise +Newsletter), or a control condition (Newsletter).
  Those exposed to the exercise intervention will have greater improvements (compared to control group) in appetite (subjective self-reported hunger responses).

SECONDARY OUTCOMES:
Assess changes in structural and functional MRI in response to an exercise intervention- prefrontal and hippocampal volume | 12 months
  Assess changes in structural and functional MRI pre- to post- intervention in sedentary youth at risk for type 2 diabetes.
  Youth randomized to the exercise intervention will exhibit increases in prefrontal and hippocampal volume compared to controls.
Assess changes in structural and functional MRI in response to an exercise intervention- reward and control | 12 months
  Assess changes in structural and functional MRI pre- to post- intervention in sedentary youth at risk for type 2 diabetes.
  Compared to pre-intervention, youth in the exercise group will show de-creased activation in reward regions (orbitofrontal cortex, ventral striatum) when making food/activity choices; increased activation in control regions (dorsolateral PFC, inferior frontal gyrus) during food/activity choices.
Assess the effectiveness of a physical activity intervention on eating behavior- subjective responses | 12 monthts
  To assess the effectiveness of a physical activity intervention on eating behavior in adolescents; OW/OB inactive adolescents will be randomly assigned to a 3-month exercise intervention (Exercise +Newsletter), or a control condition (Newsletter).
  Those exposed to the exercise intervention will have greater improvements (compared to control group) in appetite (subjective self-reported hunger responses).
Assess the effectiveness of a physical activity intervention on eating behavior- biological responses | 12 monthts
  To assess the effectiveness of a physical activity intervention on eating behavior in adolescents; OW/OB inactive adolescents will be randomly assigned to a 3-month exercise intervention (Exercise +Newsletter), or a control condition (Newsletter).
  Those exposed to the exercise intervention will have greater improvements (compared to control group) in appetite hormones ghrelin, and leptin.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Shook, PhD, Principal Investigator — Research Faculty PhD
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data will be kept private.